CLINICAL TRIAL: NCT05882019
Title: Evaluation of the "Bexa™" Breast Examination (BBE) as an Effective Solution to Breast Cancer Early Detection
Brief Title: Evaluation of the Bexa™ Breast Examination (BBE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sure, Inc. (Industry)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00067814
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 300 women presenting for screening mammograms and 400 women presenting for diagnostic mammography will undergo the Bexa Breast exam (BBE). Bexa examiners will be blinded regarding each subject's origin (screening vs. diagnostic mammogram). Each woman will receive digital breast tomosynthesis and a BBE exam on the same day. All women with a positive finding on either digital breast tomosynthesis or BBE will have an ultrasound examination of all positive findings. Up to six Bexa Certified examiners will rotate, performing the BBE's on roughly equal proportions of the subjects at a location designated within the Breast Center so as to minimally disrupt patient workflow within the site and also provide minimal inconvenience to the trial participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Breast Exam with Bexa (Other): Bexa exam to be performed on participants already scheduled for either screening or diagnostic mammography.
  Interventions: Device: Breast Exam with Bexa

INTERVENTIONS:
Device: Breast Exam with Bexa — Breast exam with Bexa uses pressure elastography to produce a map of the breast tissue's elasticity.

SUMMARY:
Objective The "Bexa Breast Exam," or "BBE," for the purposes of this study is defined as the use of a Bexa device in conjunction with a portable, focused ultrasound examination ("spot ultrasound") to identify and further evaluate abnormal breast masses including cancer. Commercially, this combination of Bexa plus focused ultrasound is called "Bexa Plus." This study compares the use of the Bexa Breast Exam (BBE/Bexa Plus) as a breast cancer early detection examination with the current standard of care digital breast tomosynthesis.

The specific objectives are:

1. To measure the sensitivity and specificity of BBE as compared to digital breast tomosynthesis.
2. Measure the proportion of women receiving a Bexa Breast Exam that require additional imaging studies.

Hypothesis The purpose of this study is to demonstrate that Bexa Breast Examination's sensitivity and specificity in identifying abnormal breast masses are equal to or superior than the standard accepted mammography with tomosynthesis.

DETAILED DESCRIPTION:
Background and Significance

Breast cancer is the second leading cause of cancer deaths among women in the United States. It is estimated that 287,850 women were diagnosed with breast cancer in 2022, of which 43,250 will die. The current recommended form of screening for breast cancer is mammography, followed by the Clinical Breast Exam, "CBE". However, CBE is subjective, highly variable depending upon training and experience, and lacks the level of sensitivity needed to consistently detect breast masses including cancer.

Mammography can be painful, irradiates the breast, is available primarily in intimidating hospital and/or medical clinic locations and requires physician interpretation. As well, screening mammography results are typically provided to the woman days to weeks after the examination. In a study of 405,191 mammogram examinations, 20% of breast cancers were missed, and 12-14% of examinations had false positives results. A study published in the February 2016 Annals of Internal Medicine posited that among women receiving annual mammography, the radiation exposure caused 246 cancers per 100,000 women over a 10-year period.

Screening mammography is not adopted by between 30% and 60% of American women over 40, with exaggerated challenges to adoption in the African American and Hispanic communities. Mammography is historically not offered to younger women, because it is inaccurate in their denser breast tissue. Over the past decade, the United States Preventive Services Task Force (USPSTF) has acted to limit the use of mammography in women 40-49 due to the high rate of false positive examinations. This has further expanded the population of women at risk for breast cancer without an effective early detection option. While annual screening remains the ideal screening frequency to achieve early detection, screening mammography recommendations from the USPSTF are driving the transition towards mammograms in women over 50 to every 24 to 36 months, primarily as a tactic to limit radiation exposure. However, this approach renders the women between the ages of 40 and 50 with no options for screening and early detection.

Globally, less than 5% of at-risk age women will ever receive screening mammography, primarily due to the expense of the equipment and of the supporting radiology operations.

Efforts must be made to improve the quality and frequency of early detection for all women at risk, particularly for those women who do not readily adhere to breast screening guidelines or for whom screening mammography is no longer a recommended option. An ideal early detection solution should be pain free, radiation free, provide immediate results, and be easily scalable to vulnerable populations. It must have both a low false negative rate and a low false positive rate, generating an acceptably low number of unnecessary referrals for additional and unneeded imaging studies. In order to make an impact upon the global community at-risk, the equipment and its operation must be low-cost, efficient, accessible and scalable. The best cancer screening test is one that patients readily adopt.

Sure, Inc. has developed a commercially available High Resolution Pressure Elastography device, the "Bexa™" device, for the detection of abnormal masses including breast cancer. The Bexa™ device uses highly accurate pressure sensors to perform elastographic evaluation of breast tissue under light compression in conjunction with proprietary image processing algorithms to identify breast masses. The device is simple to use which allows consistent results to be produced by different examiners. The Bexa™ device, hereafter referred to as "Bexa" consists of a sensor module (similar in shape to a computer mouse) with a capacitive sensor array that is connected to a tablet computer to process and visualize the results. Bexa has 510(k) clearance (K181672) from the US Food and Drug Administration (FDA) as a pressure mapping system for documentation of CBE findings under its former commercial name, "SureTouch." Sure, Inc.'s proprietary sensor array technology and processing algorithms are ideally suited for application to detection of abnormal breast masses including cancer because the technology is low-cost, highly portable, free of radiation, and consistently adopted by women in all racial and ethnic communities. Logistically, it addresses several structural and cultural barriers that prevent mass adoption of screening for breast cancer.

The Clinical Use of the Bexa Breast Exam

The majority of morbidity and mortality from breast cancer is caused by malignancies that present as solid tumors of the breast. The Bexa device produces a clear and accurate image of breast masses as small as 4mm (as measured by B-mode ultrasound) and misses between 6 and 11% of masses of all types. Mammography has a theoretical resolution of 5mm and misses 20% of breast cancers, and a higher proportion of all masses. Bexa is the best means of identifying solid masses in the breast including cancer.

In the U.S. population, Bexa will identify a mass in approximately 8%-11% of women, and these masses require additional evaluation. By comparison, mammography has a false-positive rate requiring 12%-14% of women to have unnecessary additional evaluation. The actual rate of referral for additional studies following screening mammography is often higher based upon claims review and not just false positive findings in the medical literature. As well, the literature demonstrates the known efficacy of mammography in women older than 50, with no effective solution available in the less than 50 population. Compared to mammography, the Bexa device used as an early detection technology improves mass detection accuracy while reducing the proportion of women referred for additional and unnecessary imaging studies and biopsies.

The results of the BBE are provided to women immediately whereas the results of screening mammogram examinations are require a subsequent, non-synchronous interpretation by a radiologist.

The most common next-step evaluation of a mass identified by Bexa is an ultrasound of the mass. Simple physiologic cysts and benign solid tumors can be easily identified by a focused or "spot," ultrasound of the detected mass. Based upon more than 500 masses identified by Bexa exams performed by ARDMS breast ultrasound technicians, up to half have been found to be easily identified as benign. This reduces the rate of women referred from a single visit consisting of a Bexa exam combined with "spot" ultrasound of discovered masses - which is the "Bexa Breast Exam" - to less than 4% compared to 12% -14% or more referred for additional studies following a mammogram.

The Bexa Breast Exam process produces accuracy in mass identification that exceeds the limit of lesion size and depth detectable by conventional manual palpation techniques used during a Clinical Breast Exam and digital mammography. The Bexa Breast Exam similarly requires that a far smaller proportion of women examined require additional appointments and studies compared to women undergoing mammography.

Bexa has the potential to serve as an accurate, consistent, low-cost early detection modality that can be widely deployed in U.S. and global community settings, mobile units, as well as traditional and non-traditional primary care settings.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are scheduled for a diagnostic or screening mammogram.
2. Patients of all races, ethnicities, and socio-economic background
3. Signed informed consent obtained prior to any study assessments and procedures.
4. Age 30-80 years of age and female.

Exclusion Criteria:

* Positive findings with a size in their greatest dimension > 2cm as measured by ultrasound. These masses are frequently palpable if not overtly visible and our focus, and that of other modalities used in early detection, is primarily but not exclusively the identification of non-palpable masses.
* Positive findings that cause a visible and obvious deformity of the breast or alteration in the skin appearance of the breast.
* Women with breast tenderness significant enough to prevent completion of any of the study examinations. Both ultrasound and Bexa require a light degree of pressure on the breast; certain women, very few, have enough breast tenderness that they cannot tolerate the pressure of either Bexa or ultrasound.
* Women with breast surface scarring significant enough to prevent effective BBE (keloid scarring from a previous procedure on the breast, for example).
* Greater than 3 positive findings in a given breast.
* Women who are unable to comprehend or unwilling to sign an informed consent form.
* Women ages < 30 and > 80 years of age.
* Pregnant women.
* Women who have had mastectomy - unilateral or bilateral.
* Women who have had breast cancer within the last 2 years

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 700 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Bexa sensitivity of mass detection | During procedure
  Bexa sensitivity of mass detection as compared to digital tomosynthesis mammography

SECONDARY OUTCOMES:
False Negative Comparison between Bexa and Mammography | During procedure
  Compare masses identified by one modality and missed by the other
Bexa Detected Breast Cancers | 8 weeks
  Determine how many masses detected by Bexa are biopsy-proven cancers

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cinelli, MD, Principal Investigator — Maine Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufman CS, et al., Objective measurement of the physical exam using a new device: reproducible triage of palpable masses. Breast Cancer Research and Treatment, 2004; 88; supp 1:S223-4- SABCS 2004.
- [Result] Miglioretti DL, Lange J, van den Broek JJ, Lee CI, van Ravesteyn NT, Ritley D, Kerlikowske K, Fenton JJ, Melnikow J, de Koning HJ, Hubbard RA. Radiation-Induced Breast Cancer Incidence and Mortality From Digital Mammography Screening: A Modeling Study. Ann Intern Med. 2016 Feb 16;164(4):205-14. doi: 10.7326/M15-1241. Epub 2016 Jan 12. PMID 26756460
- [Result] National Center for Health Statistics (US). Health, United States, 2016: With Chartbook on Long-term Trends in Health. Hyattsville (MD): National Center for Health Statistics (US); 2017 May. Report No.: 2017-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK453378/ PMID 28910066
- [Result] Sarvazyan A, Egorov V, Son JS, Kaufman CS. Cost-effective screening for breast cancer worldwide: current state and future directions. Breast Cancer (Auckl). 2008;1:91-9. doi: 10.4137/bcbcr.s774. Epub 2008 Jul 2. PMID 19578481
- See also: SEER 2022 — https://seer.cancer.gov/statfacts/html/breast.html
- See also: USPSTF — https://www.uspreventiveservicestaskforce.org/uspstf/recommendation/breast-cancer-screening